CLINICAL TRIAL: NCT06412913
Title: Multicenter Retrospective Observational Study to Assess the Clinical Performance and Safety Profile of MJ-FLEX in Paediatric Patients Who Have Suffered Diaphyseal Fractures of Long Bones in Daily Practice: MJ-FLEX Study
Brief Title: Retrospective Study on Clinical Performance and Safety Profile of MJ-Flex Elastic Nail
Acronym: MJ-Flex
Status: Terminated | Type: Observational
Why Stopped: This observational, retrospective study was discontinued as part of a strategic decision to reallocate resources to new product development. All patients had completed treatment before the study start.
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCI_2303; 334519 (Other: IRAS project ID (UK))
Record Dates: First submitted 2024-04-30; First posted 2024-05-14 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Fractures, Bone
Keywords: nail; elastic; elastic nailing; intramedullary; pediatric
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in pediatric age (> 18 month and < 18 years) at the time of surgery: The full analysis set includes all paediatric patients who that have been treated for diaphyseal fractures of long bones with the MJ-FLEX the will be systematically consecutive screened at the centers.
  Interventions: Device: MJ-Flex The New Metaizeau Nail

INTERVENTIONS:
Device: MJ-Flex The New Metaizeau Nail — Intramedullary implantation of the MJ-Flex elastic nail in long bones to provide bone fixation
  Other Names: Elastic Nail

SUMMARY:
This study aims to retrospectively collect data from routine clinical practice in order to evaluate the safety profile of the MJ-FLEX elastic nail used in pediatric patients according to the manufacturer Instructions For Use (IFU) in the time frame from the time of surgery until the last follow-up visit available at the hospitals.

DETAILED DESCRIPTION:
The study is planned to be conducted in two investigational sites, one in France and one in United Kingdom, both experienced in the treatment of pediatric patients with diaphyseal fractures in the clavicle and in upper and lower limbs, where the usage of MJ-Flex The New Metaizeau Nail (known as MJ-Flex) was part of the normal clinical practice.

Investigator of both study sites will provide data for a maximum of 61 patients meeting inclusion and exclusion criteria (Considering a drop-out or a non-evaluable rate of 10% of the procedures) that will contribute for approximately 61 procedures in which MJ-Flex was used.

No diagnostic or therapeutic intervention outside of routine clinical practice will be applied. The study has been designed to analyze medical records of patients where study data was collected as part of their routine clinical practice. Therefore, patients will be retrospectively enrolled in the study. Patients who have undergone MJ-Flex implantation from 02/2018 to 12/2022 are considered for the study The observation period of study subjects will comprise from surgery until the last follow up visit available.

Medical records of the participating sites are expected to contain all the required information.

In United Kingdom, no study visit will be required but according to local legislation, it will be essential that before collecting any information from medical records, participants or their guardians are asked for specific informed consent to be signed by them before any collection of patient information takes place.

However, in France, due to the use of primary data and the foreseen exemption of the informed consent (IC) form (see Section 14.2 Informed Consent), no study visit will be required.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has been adequately informed by providing the PIS. 1.1 The patient expressed his willingness to participate in the Study by signing and dating informed consent (valid only for UK patients according to local law).
2. Patients who had a regular indication for surgical intervention with MJ-Flex according to the manufacturer's IFU.
3. Patients in pediatric age (> 18 month and < 18 years) at the time of surgery.
4. Patients skeletally immature.
5. Patients who underwent surgery performed with MJ-Flex.
6. Patients with clinical data registered in her/him medical records sufficient to assess the safety and efficacy endpoint of the study: in particular, the patient has at least one follow-up at minimum 3 months from the surgery where is possible for the investigator to assess the consolidation of the treated bone.
7. The patient had surgery at least 1 year before enrollment.

Exclusion Criteria:

1. Patient who had/has a medical condition that is a contraindication according to the manufacturer's instruction for use leaflet.
2. Patient who had/has a concomitant not permitted device which cannot be safely removed.
3. Patient for whom there are other concurrent medical or other conditions that in the opinion of the participating investigator may prevent participation or otherwise render the patient ineligible for the study.
4. The patient had surgery less than 1 year before enrollment.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The full analysis set includes all paediatric patients who that have been treated for diaphyseal fractures of long bones with the MJ-FLEX the will be systematically consecutive screened at the centers.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Percentage of procedures that have achieved bone union at the "bone consolidation assessment" visit | After 5 month (approximately) from surgery
  The measurement of efficacy will be mande with the percentage of procedures that have achieved bone union
Percentage of procedures with at least one serious/not serious adverse event certainly related or possibly related to MJ-FLEX (ADEs/SADEs) | from the date of surgery until the last follow-up, assessed up to 1 year
  This outcome will be used to measure safety
Percentage of procedures who experienced at least one MDDs that caused an effect on the patient | from the date of surgery until the last follow-up, assessed up to 1 year
  This outcome will be used to measure safety
Post-treatment fracture-free survival | up to 1 year
  This outcome will be used to measure safety

CONTACTS AND LOCATIONS:
Overall Officials: Sara Dorman, MD, Principal Investigator — Sheffield Children's NHS Foundation Trust
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No